CLINICAL TRIAL: NCT04228783
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Immunogenicity, Safety, Reactogenicity, and Consistency of a Heterologous 2-dose Vaccine Regimen Using 3 Consecutive Lots of Ad26.ZEBOV and MVA-BN®-Filo in Adult Participants
Brief Title: A Study of 2-dose Vaccine Regimen Using 3 Consecutive Lots of Ad26.ZEBOV and MVA-BN-Filo in Adult Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108694; VAC52150EBL3004 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Ebola
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Active Vaccine: Group 1 (Ad26.ZEBOV-Lot A, MVA-BN-Filo-Lot 1) (Experimental): Participants will receive Intramuscular injection (0.5 milliliter [mL]) of Adenovirus serotype 26 encoding the Ebola virus Mayinga glycoprotein (Ad26.ZEBOV) as Dose 1 (5*10^10 viral particle(s) [vp], Lot A) on Day 1, followed by Modified Vaccinia Ankara Bavarian Nordic vector encoding multiple filovirus proteins (MVA-BN-Filo) as Dose 2 (1*10^8 infectious unit(s) [Inf U], Lot 1) on Day 57.
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo
- Active Vaccine: Group 2 (Ad26.ZEBOV-Lot B, MVA-BN-Filo-Lot 2) (Experimental): Participants will receive Intramuscular injection (0.5 mL) of Ad26.ZEBOV as Dose 1 (5*10^10 vp, Lot B) on Day 1, followed by MVA-BN-Filo as Dose 2 (1*10^8 Inf U, Lot 2) on Day 57.
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo
- Active Vaccine: Group 3 (Ad26.ZEBOV-Lot C, MVA-BN-Filo-Lot 3) (Experimental): Participants will receive Intramuscular injection (0.5 mL) of Ad26.ZEBOV as Dose 1 (5*10^10 vp, Lot C) on Day 1, followed by MVA-BN-Filo as Dose 2 (1*10^8 Inf U, Lot 3) on Day 57.
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo
- Control Vaccine: Group 4 (Placebo) (Placebo Comparator): Participants will receive Intramuscular injection (0.5 mL) of placebo (0.9 percent [%] saline) matching to Ad26.ZEBOV as Dose 1 on Day 1, followed by placebo matching to MVA-BN-Filo as Dose 2 on Day 57.
  Interventions: Biological: Placebo
- Booster Cohort: Group 5 (Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV) (Experimental): Participants will receive Intramuscular injection (0.5 mL) of Ad26.ZEBOV as Dose 1 (5*10^10 vp, a single Lot) on Day 1, followed by MVA-BN-Filo as Dose 2 (1*10^8 Inf U, a single Lot) on Day 57 and a booster dose of Ad26.ZEBOV (at a dose of 5*10^10 vp, a single Lot) 4 months after Dose 2 (on Day 177).
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo
- Booster Cohort: Group 6 (Placebo) (Placebo Comparator): Participants will receive Intramuscular injection (0.5 mL) of placebo (0.9% saline) matching to Ad26.ZEBOV as Dose 1 on Day 1, followed by placebo matching to MVA-BN-Filo as Dose 2 on Day 57 and a booster dose of matching placebo on Day 177.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ad26.ZEBOV — Participants will receive IM injection (0.5 mL) of Ad26.ZEBOV as Dose 1 (5*10^10 vp, Lot A, B, and C) on Day 1 (Groups 1, 2, 3 and 5) and an Ad26.ZEBOV booster dose on Day 177 (Group 5).
  Arms: Active Vaccine: Group 1 (Ad26.ZEBOV-Lot A, MVA-BN-Filo-Lot 1); Active Vaccine: Group 2 (Ad26.ZEBOV-Lot B, MVA-BN-Filo-Lot 2); Active Vaccine: Group 3 (Ad26.ZEBOV-Lot C, MVA-BN-Filo-Lot 3); Booster Cohort: Group 5 (Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV)
Biological: MVA-BN-Filo — Participants will receive IM injection (0.5 mL) of MVA-BN-Filo as Dose 2 (1*10^8 Inf U, Lot 1, 2, 3 and 5) on Day 57.
  Arms: Active Vaccine: Group 1 (Ad26.ZEBOV-Lot A, MVA-BN-Filo-Lot 1); Active Vaccine: Group 2 (Ad26.ZEBOV-Lot B, MVA-BN-Filo-Lot 2); Active Vaccine: Group 3 (Ad26.ZEBOV-Lot C, MVA-BN-Filo-Lot 3); Booster Cohort: Group 5 (Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV)
Biological: Placebo — Participants will receive IM injection (0.5 mL) of placebo (0.9 % saline) as Dose 1 on Day 1, followed by placebo as Dose 2 on Day 57 (Groups 4 and 6) and a booster of matching placebo on Day 177 (Group 6).
  Arms: Booster Cohort: Group 6 (Placebo); Control Vaccine: Group 4 (Placebo)

SUMMARY:
The purpose of this study is to demonstrate that the paired 2-dose vaccine regimens from 3 consecutively manufactured lots of Adenovirus serotype 26 encoding the Ebola virus Mayinga glycoprotein (Ad26.ZEBOV) as Dose 1 and 3 consecutively manufactured lots of Modified Vaccinia Ankara Bavarian Nordic vector encoding multiple filovirus proteins (MVA-BN-Filo) including the ebola virus mayinga glycoprotein as Dose 2, administered at a 56-day interval, induce an equivalent humoral immune response.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent form (ICF)
* Medically stable in the investigator's clinical judgment on the basis of physical examination, medical history, and vital signs performed at screening
* Before randomization, a woman must be either: a. Not of childbearing potential; b. Of childbearing potential and practicing an acceptable effective method of birth control and agrees to remain on such a method of birth control from signing the informed consent form (ICF) until at least 3 months post Dose 1 vaccination or 28 days post Dose 2 vaccination or 3 months post booster vaccination (Groups 5-6 only), whichever comes later. Use of hormonal contraception should start at least 28 days before the first administration of study vaccine. Acceptable effective methods for this study include: 1) hormonal contraception; 2) intrauterine device (IUD); 3) intrauterine hormone-releasing system (IUS); 4) male or female condom with or without spermicide; 5) cap, diaphragm, or sponge with a vaginal spermicide; 6) vasectomized partner (the vasectomized partner should be the sole partner for that participant); 7) sexual abstinence
* Women of childbearing potential must have a negative urine Beta-human chorionic gonadotropin (Beta-hCG) pregnancy test at screening and immediately prior to each study vaccine administration
* Available and willing to participate for the duration of the study and follow-up visit
* Willing to provide verifiable identification

Exclusion Criteria:

* Having received any candidate Ebola vaccine
* Diagnosed with Ebola virus disease (EVD), or prior exposure to Ebola virus, including travel to an area with Ebola outbreak less than 1 month prior to screening (if applicable)
* Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines), including known allergy to egg, egg products, and aminoglycosides
* Presence of acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature greater than or equal to (>=) 38.0ºCelcius on Day 1. Participants with such symptoms will be excluded from enrollment at that time but may be rescheduled for enrollment at a later date
* Human immunodeficiency virus (HIV) type 1 or type 2 infection, based on the medical history reported by the participant
* Pregnant, breast-feeding
* History of an underlying clinically significant acute or chronic medical condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 974 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (7):
- United States (7):
  - Coastal Clinical Research, Inc, Mobile, Alabama
  - Clinical Research Consortium, an AMR company, Tempe, Arizona
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - The Center For Pharmaceutical Research, Kansas City, Missouri
  - Clinical Research Consortium, an AMR company, Las Vegas, Nevada
  - AMR New Orleans, Formerly New Orleans Center for Clinical Research - New Orleans, an AMR company, Knoxville, Tennessee
  - Alliance for Multispeciality Research, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 974 participants were enrolled and randomized, of which 970 participants received the vaccination and were included in the analysis.
Groups:
- Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1): Participants received 0.5 milliliter (mL) intramuscular injection of adenovirus serotype 26 encoding the Ebola virus Mayinga glycoprotein (Ad26.ZEBOV) as Dose 1 (5*10^10 viral particles [vp], Lot A) on Day 1, followed by intramuscular injection of modified vaccinia Ankara Bavarian Nordic vector encoding multiple filovirus proteins (MVA-BN-Filo) as Dose 2 (1*10^8 infectious units [Inf U], Lot 1) on Day 57.
- Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2): Participants received 0.5 mL intramuscular injection of Ad26.ZEBOV as Dose 1 (5*10^10 vp, Lot B) on Day 1, followed by intramuscular injection of MVA-BN-Filo as Dose 2 (1*10^8 Inf U, Lot 2) on Day 57.
- Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3): Participants received 0.5 mL intramuscular injection of Ad26.ZEBOV as Dose 1 (5*10^10 vp, Lot C) on Day 1, followed by intramuscular injection of MVA-BN-Filo as Dose 2 (1*10^8 Inf U, Lot 3) on Day 57.
- Placebo, Placebo (Group 4): Participants received 0.5 mL intramuscular injection of placebo (0.9 percent [%] saline) matching to Ad26.ZEBOV as Dose 1 on Day 1, followed by intramuscular injection of placebo matching to MVA-BN-Filo as Dose 2 on Day 57.
- Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV (Group 5): Participants received 0.5 mL intramuscular injection of Ad26.ZEBOV as Dose 1 (5*10^10 vp, a single Lot) on Day 1, followed by intramuscular injection of MVA-BN-Filo as Dose 2 (1*10^8 Inf U, a single Lot) on Day 57 and an intramuscular injection of booster dose of Ad26.ZEBOV (at a dose of 5*10^10 vp, a single Lot) 4 months after Dose 2 (on Day 177).
- Placebo, Placebo, Placebo (Group 6): Participants received 0.5 mL intramuscular injection of placebo (0.9% saline) matching to Ad26.ZEBOV as Dose 1 on Day 1, followed by intramuscular injection of placebo matching to MVA-BN-Filo as Dose 2 on Day 57, and intramuscular injection of placebo matching to Ad26.ZEBOV booster on Day 177.
Period: Overall Study
Arm/Group | Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) | Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2) | Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3) | Placebo, Placebo (Group 4) | Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV (Group 5) | Placebo, Placebo, Placebo (Group 6)
Started | 287 | 288 | 287 | 48 | 50 | 10
Completed | 239 | 237 | 236 | 39 | 33 | 6
Not Completed | 48 | 51 | 51 | 9 | 17 | 4
Not completed — Adverse Event | 1 | 0 | 2 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 36 | 36 | 28 | 6 | 14 | 3
Not completed — Physician Decision | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 10 | 19 | 1 | 2 | 0
Not completed — Other | 4 | 3 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) | Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2) | Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3) | Placebo, Placebo (Group 4) | Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV (Group 5) | Placebo, Placebo, Placebo (Group 6) | Total
Number analyzed (Participants) | 287 | 288 | 287 | 48 | 50 | 10 | 970
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (9.32) | 34.7 (9.12) | 35.3 (8.96) | 35 (8.66) | 32.5 (7.26) | 35 (7.83) | 35 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 159 | 158 | 25 | 29 | 4 | 534
  Male | 128 | 129 | 129 | 23 | 21 | 6 | 436
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 25 | 16 | 4 | 0 | 0 | 76
  Not Hispanic or Latino | 256 | 260 | 270 | 44 | 50 | 10 | 890
  Unknown or Not Reported | 0 | 3 | 1 | 0 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 4 | 0 | 1 | 0 | 10
  Asian | 3 | 6 | 8 | 0 | 0 | 0 | 17
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 2 | 0 | 0 | 0 | 5
  Black or African American | 77 | 87 | 78 | 21 | 19 | 5 | 287
  White | 198 | 185 | 185 | 26 | 30 | 5 | 629
  More than one race | 3 | 6 | 10 | 0 | 0 | 0 | 19
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 0 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 287 | 288 | 287 | 48 | 50 | 10 | 970

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentrations (GMCs) of Binding Antibody Levels Against the Ebola Virus Glycoprotein (EBOV GP) as Measured by Enzyme-linked Immunosorbent Assay (ELISA) at 21 Days Post Vaccination 2
Description: Antibody GMCs against the EBOV GP as measured by ELISA at 21 days post Vaccination 2 were reported. GMCs of antibodies binding to EBOV GP using ELISA were reported and were measured in ELISA units per milliliter (EU/mL). Serum samples were collected for analysis of binding antibodies against EBOV GP using ELISA to determine humoral responses following vaccination. For ELISA binding antibody responses, values below the lower limit of quantification (LLOQ) of 36.11 EU/mL were imputed with half of the LLOQ prior to the computation of the GMCs.
Time Frame: 21 Days Post Vaccination 2 (Day 78)
Population: Per protocol (PP) analysis set included all randomized (Group 1-4 only) and vaccinated participants, who received Dose 1 and Dose 2 vaccinations, and booster vaccination (Groups 5 and 6 only) (administered within protocol-defined window), had at least 1 post vaccination (after date of vaccination) evaluable immunogenicity sample, had no major protocol deviations influencing the immune response. N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) | Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2) | Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3) | Placebo, Placebo (Group 4) | Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV (Group 5) | Placebo, Placebo, Placebo (Group 6)
Number analyzed (Participants) | 163 | 163 | 149 | 27 | 34 | 4
EU/mL | 11077 [9806 to 12514] | 12223 [10665 to 14010] | 11818 [10320 to 13534] | NA [NA to NA] — Here, 'NA' signifies that geometric mean and lower and upper limit of 95% CI was less than LLOQ. | 18877 [14173 to 25142] | NA [NA to NA] — Here, 'NA' signifies that geometric mean and lower and upper limit of 95% CI was less than LLOQ.
Statistical Analysis 1: Comparison: Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) vs Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2); Test type: Equivalence — An equivalence margin of 0.5 to 2.0 was considered relevant to demonstrate the equivalence of the two products; Ratio of GMCs = 0.9, 95% CI 2-sided [0.8 to 1.1]
Statistical Analysis 2: Comparison: Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) vs Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3); Test type: Equivalence — An equivalence margin of 0.5 to 2.0 was considered relevant to demonstrate the equivalence of the two products; Ratio of GMCs = 0.9, 95% CI 2-sided [0.8 to 1.1]
Statistical Analysis 3: Comparison: Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2) vs Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3); Test type: Equivalence — An equivalence margin of 0.5 to 2.0 was considered relevant to demonstrate the equivalence of the two products; Ratio of GMCs = 1.0, 95% CI 2-sided [0.9 to 1.2]

2. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Binding Antibody Levels Against the Ebola Virus Glycoprotein (EBOV GP) as Measured by Enzyme-linked Immunosorbent Assay (ELISA) at 56 Days Post Vaccination 1
Description: Antibody GMCs against the EBOV GP as measured by ELISA at 56 days post Vaccination 1 were reported. GMCs of antibodies binding to EBOV GP using ELISA were reported and were measured in ELISA units per milliliter (EU/mL). Serum samples were collected for analysis of binding antibodies against EBOV GP using ELISA to determine humoral responses following vaccination. For ELISA binding antibody responses, values below the LLOQ of 36.11 EU/mL were imputed with half of the LLOQ prior to the computation of the GMCs.
Time Frame: 56 Days Post Vaccination 1 (Day 57)
Population: PP analysis set included all randomized (Groups 1-4 only) and vaccinated participants, who received Dose 1 and Dose 2 vaccinations, and booster vaccination (Groups 5 and 6 only) (administered within protocol-defined window), had at least 1 post vaccination (after date of vaccination) evaluable immunogenicity sample, had no major protocol deviations influence the immune response. Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) | Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2) | Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3) | Placebo, Placebo (Group 4) | Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV (Group 5) | Placebo, Placebo, Placebo (Group 6)
Number analyzed (Participants) | 175 | 177 | 166 | 29 | 39 | 6
EU/mL | 988 [842 to 1159] | 994 [865 to 1142] | 960 [819 to 1126] | NA [NA to NA] — Here, 'NA' signifies that geometric mean and lower and upper limit of 95% CI was less than LLOQ. | 1023 [773 to 1354] | NA [NA to 37] — Here, 'NA' signifies that geometric mean and lower limit of 95% CI was less than LLOQ.
Statistical Analysis 1: Comparison: Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) vs Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2); Test type: Equivalence — An equivalence margin of 0.5 to 2.0 was considered relevant to demonstrate the equivalence of the two products; Ratio of GMCs = 1.0, 95% CI 2-sided [0.8 to 1.2]
Statistical Analysis 2: Comparison: Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) vs Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3); Test type: Equivalence — An equivalence margin of 0.5 to 2.0 was considered relevant to demonstrate the equivalence of the two products; Ratio of GMCs = 1.0, 95% CI 2-sided [0.8 to 1.3]
Statistical Analysis 3: Comparison: Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2) vs Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3); Test type: Equivalence — An equivalence margin of 0.5 to 2.0 was considered relevant to demonstrate the equivalence of the two products; Ratio of GMCs = 1.0, 95% CI 2-sided [0.8 to 1.3]

3. Secondary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) Until 7 Days After Vaccination 1 and 2
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their diary for 7 days post vaccination. Solicited local AEs were injection site pain/tenderness, erythema, induration/swelling, itching, pruritis at the vaccination site.
Time Frame: Until 7 Days after Vaccination 1 on Day 1 (Up to Day 8); Until 7 Days after Vaccination 2 on Day 57 (Up to Day 64)
Population: Full analysis set (FAS) included all participants with at least one study vaccine administration documented. Here, "n (number analyzed)" signifies number of participants who were analyzed at the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) | Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2) | Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3) | Placebo, Placebo (Group 4) | Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV (Group 5) | Placebo, Placebo, Placebo (Group 6)
Number analyzed (Participants) | 287 | 288 | 287 | 48 | 50 | 10
Participants
  Until 7 days after Vaccination 1 | 169 | 176 | 178 | 11 | 38 | 2
  Until 7 days after Vaccination 2: number analyzed (Participants) | 253 | 253 | 250 | 43 | 49 | 8
  Until 7 days after Vaccination 2 | 95 | 107 | 106 | 11 | 21 | 2

4. Secondary Outcome: Number of Participants With Solicited Systemic Adverse Events (AEs) Until 7 Days After Vaccination 1 and 2
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. Participants recorded the temperature in the e-Diary in the evening of the day of vaccination, and then daily for the next 7 days approximately at the same time each day. If more than 1 measurement was made on any given day, the highest temperature of that day was recorded in the e-Diary. Fever was defined as endogenous elevation of body temperature greater than or equal to (>=) 38.0 degree Celsius or >=100.4-degree Fahrenheit, as recorded in at least 1 measurement. Participants also noted the signs and symptoms in the e-Diary on a daily basis for 7 days post vaccination 1 and 2 (day of vaccination and the subsequent 7 days), if feasible, for the following events: fatigue, headache, nausea, myalgia, arthralgia, chills, and fever.
Time Frame: Until 7 Days after Vaccination 1 on Day 1 (Up to Day 8); Until 7 Days after Vaccination 2 on Day 57 (Up to Day 64)
Population: FAS included all participants with at least one study vaccine administration documented. Here, "n (number analyzed)" signifies number of participants who were analyzed at the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) | Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2) | Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3) | Placebo, Placebo (Group 4) | Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV (Group 5) | Placebo, Placebo, Placebo (Group 6)
Number analyzed (Participants) | 287 | 288 | 287 | 48 | 50 | 10
Participants
  Until 7 days after Vaccination 1 | 162 | 144 | 156 | 18 | 37 | 2
  Until 7 days after Vaccination 2: number analyzed (Participants) | 253 | 253 | 250 | 43 | 49 | 8
  Until 7 days after Vaccination 2 | 74 | 90 | 95 | 14 | 19 | 3

5. Secondary Outcome: Number of Participants With Unsolicited Adverse Events (AEs) Until 28 Days After Vaccination 1 and 2
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. Unsolicited AEs were all AEs for which the participant was not specifically questioned in the participant diary.
Time Frame: Until 28 Days After Vaccination 1 on Day 1 (Up to Day 29); until 28 days after Vaccination 2 on Day 57 (Up to Day 85)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) | Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2) | Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3) | Placebo, Placebo (Group 4) | Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV (Group 5) | Placebo, Placebo, Placebo (Group 6)
Number analyzed (Participants) | 287 | 288 | 287 | 48 | 50 | 10
Participants
  Until 28 days after Vaccination 1 | 28 | 25 | 26 | 0 | 1 | 1
  Until 28 days after Vaccination 2: number analyzed (Participants) | 253 | 253 | 250 | 43 | 49 | 8
  Until 28 days after Vaccination 2 | 14 | 8 | 17 | 3 | 0 | 0

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAE was any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Day 1 up to Day 237 for Groups 1, 2, 3, 4, and up to Day 537 for Groups 5 and 6
Population: FAS included all participants with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) | Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2) | Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3) | Placebo, Placebo (Group 4) | Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV (Group 5) | Placebo, Placebo, Placebo (Group 6)
Number analyzed (Participants) | 287 | 288 | 287 | 48 | 50 | 10
Participants | 4 | 1 | 6 | 1 | 3 | 1

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 237 for Groups 1, 2, 3, 4, and up to Day 537 for Groups 5 and 6
Description: Full analysis set (FAS) included all participants with at least one study vaccine administration documented.
Arm/Group | Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) | Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2) | Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3) | Placebo, Placebo (Group 4) | Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV (Group 5) | Placebo, Placebo, Placebo (Group 6)
All-Cause Mortality (participants affected / at risk) | 0/287 | 0/288 | 0/287 | 0/48 | 1/50 | 0/10
Serious Adverse Events (participants affected / at risk) | 4/287 | 1/288 | 6/287 | 1/48 | 3/50 | 1/10
Other Adverse Events (participants affected / at risk) | 0/287 | 0/288 | 0/287 | 0/48 | 2/50 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) (N=287) | Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2) (N=288) | Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3) (N=287) | Placebo, Placebo (Group 4) (N=48) | Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV (Group 5) (N=50) | Placebo, Placebo, Placebo (Group 6) (N=10)
Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Ophthalmic Herpes Zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Fracture Displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Stab Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Venomous Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alcoholic Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 1
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Accelerated Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ad26.ZEBOV(Lot A), MVA-BN-Filo (Lot 1) (Group 1) (N=287) | Ad26.ZEBOV(Lot B), MVA-BN-Filo (Lot 2) (Group 2) (N=288) | Ad26.ZEBOV(Lot C), MVA-BN-Filo (Lot 3) (Group 3) (N=287) | Placebo, Placebo (Group 4) (N=48) | Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV (Group 5) (N=50) | Placebo, Placebo, Placebo (Group 6) (N=10)
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT04228783/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT04228783/SAP_001.pdf